## Comparison of Standard PET/CT Versus Digital PET/CT

NCT03081767

March 16, 2022

Andrei Iagaru, Principal Investigator Stanford University Stanford, California 94305

Statistical Analysis Plan

Image quality was evaluated using a 5-point Likert scale: 5 - Diagnostic: Excellent diagnostic image quality; 4 - Diagnostic: Good diagnostic image quality; 3 - Diagnostic: Acceptable diagnostic image quality; 2 - Sub-optimal diagnostic: image quality with limited additional clinical information; 1 - Non-diagnostic: non-diagnostic image quality. Statistical analysis was performed with Microsoft Excel for Mac version 16.58 (Microsoft Corporation, Redmond, WA, USA).

Continuous data are presented as mean  $\pm$  standard deviation (SD), minimum (min) - maximum (max) values. A two-tailed, paired Student's T-Test was used to assess significance in Likert score between the standard and digital PET/CT scanner. A P-value of <0.05 was considered significant.